CLINICAL TRIAL: NCT02389075
Title: The Colonic Microbiome and Mucosal Immunity in Inflammatory Bowel Disease and Ankylosing Spondylitis
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-1507; UL1TR001082 (NIH)
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Bowel Diseases (IBD); Ankylosing Spondylitis (AS)
Keywords: intraepithelial lymphocytes (IEL); microbiome; colon mucosa
MeSH Terms: conditions — Inflammatory Bowel Diseases; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Colon pinch biopsies, white blood cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ankylosing Spondylitis: Subjects with a diagnosis of ankylosing spondylitis undergoing routine colonoscopy or willing to undergo a flexible sigmoidoscopy for research purposes only. They will be asked to fill out questionnaires, give blood, perform a rectal swab, and have pinch biopsies taken during endoscopy.
  Interventions: Procedure: Pinch biopsies; Procedure: Flexible sigmoidoscopy
- Inflammatory Bowel Disease: Subjects with a diagnosis of inflammatory bowel disease undergoing routine colonoscopy. They will be asked to fill out questionnaires, give blood, perform a rectal swab, and have pinch biopsies taken during endoscopy.
  Interventions: Procedure: Pinch biopsies
- Healthy Controls: Subjects without any major autoimmune diseases or pathologies undergoing routine colonoscopy. They will be asked to fill out questionnaires, give blood, perform a rectal swab, and have pinch biopsies taken during endoscopy.
  Interventions: Procedure: Pinch biopsies

INTERVENTIONS:
Procedure: Pinch biopsies — Biopsies obtained during colonoscopy or flexible sigmoidoscopy.
Procedure: Flexible sigmoidoscopy — Offered to subjects with ankylosing spondylitis who do not meet criteria for colonoscopy
  Groups: Ankylosing Spondylitis

SUMMARY:
This study plans to learn more about the relationship between systemic autoimmune disease, such as inflammatory bowel disease and ankylosing spondyloarthritis, bacteria in the colon, and the changes in colon tissue.

DETAILED DESCRIPTION:
Changes in human gut bacteria has been shown in patients with autoimmune diseases, such as inflammatory bowel diseases (IBD). The gut flora in ankylosing spondylitis (AS), an arthritis that can occur with IBD, has not been well studied. The immune cells in the colon directly interface with bacteria and may be influenced by them. The interactions between the colon immune system, bacteria and autoimmunity hasn't been studied. The study goal is to specifically study the link between bacteria, the colonic immune system, and the autoimmune diseases of AS and IBD. This will be done by collecting clinical data by questionnaires, blood samples, colonic tissue during endoscopy, and microbiome data in subjects with IBD, AS, and controls.

ELIGIBILITY:
Healthy Controls

Exclusion criteria:

* Pregnancy
* Use of antibiotics within the past 14 days†
* Current diagnosis of colon cancer
* Diagnosis of celiac disease
* Diagnosis of any other rheumatologic disease such as RA, SLE, etc.
* Chemotherapy or radiation therapy for any malignancy within the past year
* Daily use of aspirin or NSAIDs with inability to hold the drug 7 days before and after the procedure
* Current use of anticoagulation (LMWH,warfarin,etc.)
* A diagnosis of HIV
* Clostridium difficile within the past 3 months

IBD

Inclusion Criteria:

* Established IBD (either Crohn's disease or ulcerative colitis)
* Suspected to have IBD by a gastroenterologist and undergoing diagnostic endoscopy and biopsy. Diagnosis will be confirmed on biopsy and patients who are negative will be considered for controls based on the pathology found.

Exclusion Criteria:

* Pregnancy
* Use of antibiotics within the past 14 days
* Current diagnosis of colon cancer
* Diagnosis of celiac disease
* Diagnosis of any other rheumatologic disease such as RA, SLE, etc.
* Chemotherapy or radiation therapy for any malignancy within the past year
* Daily use of aspirin or NSAIDs with inability to hold the drug 7 days before and after the procedure
* Current use of anticoagulation (LMWH, warfarin,etc.)
* A diagnosis of HIV
* Clostridium difficile within the past 3 months
* Evidence of inflammatory spinal or axial arthritis or disease based on chart review such as inflammation seen on radiographs or a diagnosis of sacroiliitis

AS:

Inclusion Criteria:

* Diagnosed with an axial spondyloarthritis (SpA) by a rheumatologist -
* Meet the Assessment of SpondyloArthritis international Society (ASAS) axial spondyloarthritis (SpA) criteria

Exclusion criteria:

* Pregnancy
* Use of antibiotics within the past 14 days
* Current diagnosis of colon cancer
* Diagnosis of celiac disease
* Diagnosis of any other rheumatologic disease such as RA, SLE, etc.
* Chemotherapy or radiation therapy for any malignancy within the past year
* Daily use of aspirin or NSAIDs with inability to hold the drug 7 days before and after the procedure
* Current use of anticoagulation (LMWH,warfarin,etc.)
* A diagnosis of HIV
* Clostridium difficile within the past 3 months
* A known history of idiopathic macroscopic or microscopic colitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inflammatory Bowel Disease, Ankylosing Spondylitis, and Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2015-03; Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
IEL characteristics in IBD, AS, and healthy controls | 1 hour after colonoscopy
  The primary goal for this measure will be to demonstrate characteristics of IEL (intraepithelial lymphocytes) subtypes of healthy individuals and compare those with AS or IBD. IEL characteristics will be based on cell marker outcomes using flow cytometry for CD3, CD4, CD8α, CD8β, CD44, CD45, CD62L, CD69, CD103, TCRαβ, and TCRγδ.

SECONDARY OUTCOMES:
Microbiome Differences in IBD, AS, and healthy controls | 1 hour after colonoscopy
  The primary hypothesis is that the microbiome population will differ between controls, IBD, and AS; outcomes for this hypothesis will include relative abundance (RA) of individual bacterial species and the Shannon Index for community diversity.
Microbiome changes are reflected in IELs | 1 hour after colonoscopy
  The primary hypothesis is that dysbiosis will be reflected in the IEL populations in AS and IBD by having a different predominant phenotype (as seen by cell markers) compared to healthy controls; the investigators will evaluate the IEL outcomes determined to be significantly different among AS, IBD, and healthy controls as identified in Outcome 1 (Primary Outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Kuhn, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Regner EH, Ohri N, Stahly A, Gerich ME, Fennimore BP, Ir D, Jubair WK, Gorg C, Siebert J, Robertson CE, Caplan L, Frank DN, Kuhn KA. Functional intraepithelial lymphocyte changes in inflammatory bowel disease and spondyloarthritis have disease specific correlations with intestinal microbiota. Arthritis Res Ther. 2018 Jul 20;20(1):149. doi: 10.1186/s13075-018-1639-3. PMID 30029674